CLINICAL TRIAL: NCT04133285
Title: Registry of Multiple Osteochondromas That Collects Clinical, Functional, Genetic, Genealogical, Imaging, Surgical, Treatment, Quality of Life Data. Data is Linked to Patients' Biological Samples, When Available.
Brief Title: Registry of Multiple Osteochondromas
Acronym: REM
Status: Recruiting | Type: Observational
Sponsor: Luca Sangiorgi (Other)
Responsible Party: Sponsor-Investigator, Luca Sangiorgi, Head of Department of Rare Skeletal Disorders, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: 21629/2013
Record Dates: First submitted 2019-10-14; First posted 2019-10-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Multiple Osteochondromas
Keywords: Disease Registry; Natural History Study; Disease evolution; Genotype-Phenotype Correlation
MeSH Terms: conditions — Exostoses, Multiple Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples With DNA — Whole peripheral blood, DNA, lymphocytes, cartilage tissues, bone tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Osteochondromas patients: Patients affected by Multiple Osteochondromas. The Registry will include also data on fetuses (prenatal).

SUMMARY:
REM is a retrospective and prospective registry, finalized for care and research purposes. It is articulated in main sections - strongly related and mutually dependent on each other - corresponding to different data domains: personal information, clinical data, genetic data, genealogical data, surgeries, etc.

This approach has been developed to corroborate and integrate data from different sources evaluating several aspects of diseases and to correlate genetic background and phenotypic outcomes, in order to better investigate disease pathophysiology. Due to legal requirements, institutional directives and organizational issues, we are unable to include individuals residing outside Italy in the registry at this time. We are currently engaged in the preparation of a recruitment process for individuals residing outside Italy.

DETAILED DESCRIPTION:
The traditional method of collecting patient information is often chaotic, inconvenient, and sometimes even unsafe, particularly when dealing with rare diseases. In 2013, the need to simplify the diagnostic process and to overcome the difficulties of data storage and analysis, led to the suggestion of implementing the Registry of Multiple Osteochondromas (REM).

The REM relies on an IT platform named Genotype-phenotype Data Integration platform - GeDI. This solution was developed through a collaboration between Rare Skeletal Disease Department and a local software company (Dilaxia S.p.A.) and is General Data Protection Regulation (GDPR)-compliant, multi-client and web-accessible. It has been designed according to current medical informatics standards, including the Orphanet code, the International Classification of Diseases (ICD), and the Human Genome Variants Society, aiming to follow Findability, Accessibility, Interoperability, Reusability (FAIR) principles. GeDI is continuously being implemented to improve the management of people with Multiple Osteochondromas and to assist researchers in analyzing the information collected. REM is divided into the following main sections:

* Personal data: it comprises general information, birth details and residence data;
* Patient data: including the patients internal code, the hospital code and other patient details;
* Diagnostic Process: the diagnosis, the status (affected, suspected, etc.), age at diagnosis, comorbidities, allergies, etc.;
* Genogram: a tool for designing the family transmission of the disease, alongside information on the disease status of all relatives included;
* Clinical events: it records a long list of signs and symptoms of Multiple Osteochondromas as well as several additional items to describe the disease
* Genetic Analysis and Alteration: including analytical technique, sample information, analysis duration, etc. This section also comprises detailed information on any detected pathological variants (e.g. gene, international reference, DNA change, protein change, genomic position, etc.);
* Visits: this section includes visit type (genetic, orthopedic, rehabilitation, pediatric, etc.), the date of the visit, prescriptions, imaging, etc.;
* Treatments: this section comprises information of a wide range of treatments including pharmacological, devices, supplements, and other treatments such as psychological, nutritional, etc;
* Surgeries: this section contains information on the type of surgeries, the age of the patients, the site/localization of the procedures, etc.
* Documents: this repository allow us to store all types of documents (radiological reports, imaging, consents, clinical reports, etc.);
* Consents: this section provides a comprehensive overview of all consents collected, including the collection date;
* Samples: this section includes information on the samples, like the type, date of collection, etc.
* PROs: this section collects information on patients reported outcomes such as the quality of life or ABC scale.

ELIGIBILITY:
Inclusion Criteria:

* All Multiple Osteochondromas patients, including prenatal diagnosis of Multiple Osteochondromas

Exclusion Criteria:

* Any condition unrelated to Multiple Osteochondromas

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by Multiple Osteochondromas. The Registry will include also data on fetuses (prenatal).
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-06-28 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Natural History and Epidemiology in terms of clinical, genetic and functional evaluation | 25 years
  To maintain an established registry in order to assess epidemiology and natural history.
  Collection of:
  1. physical examinations data: assessment of severity of the disease (according to Mordenti et al classification)
  2. orthopedic and functional data: stature (cm), weight (kg), number and localization of sites affected, site of malignant transformation, definition of deformities (localization and number), definition of limitations (localization and number)
  3. surgical procedures: type, number and site of surgeries disease-related and age at surgeries
  4. genetics background: target gene, type of mutation, type of variant detected, clinical significance
  5. family history: inheritance
  6. treatment information: pharmacological, devices, supplements, and other treatments
  All the features are updated at each follow up. Clinical reports, medical charts, genetic report and imaging are the primary sources of data

SECONDARY OUTCOMES:
Genotype-Phenotype Correlation among clinical features and molecular background | 25 years
  The secondary outcome comprises the correlation between genotype and phenotype. This includes but is not limited to clinical features and genetic background. This will be pursued using the information collected during visits and follow-ups and the genetic information resulting from molecular investigations.

OTHER OUTCOMES:
Longitudinal study of disease evolution (including prospective and retrospective data) | 25 years
  This outcome aims to investigate the evolution of Multiple Osteochondromas during time. This will be evaluated within the families and among the families.
  Main clinical features, such as height (cm), number and localization of osteochondromas, number and localization of deformities, number and localization of limitations will be collected both retrospectively and prospectively in the entire population, with a particular attention to the pediatric population. Primarily in adult population, disease evolution is focused on malignant transformation. An evaluation of these parameters will be performed at each visit to keep track on the progression of clinical manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Sangiorgi, MD, PhD, MS, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Irccs Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

REFERENCES:
- [Background] Mordenti M, Ferrari E, Pedrini E, Fabbri N, Campanacci L, Muselli M, Sangiorgi L. Validation of a new multiple osteochondromas classification through Switching Neural Networks. Am J Med Genet A. 2013 Mar;161A(3):556-60. doi: 10.1002/ajmg.a.35819. Epub 2013 Feb 8. PMID 23401177
- [Background] Pedrini E, Jennes I, Tremosini M, Milanesi A, Mordenti M, Parra A, Sgariglia F, Zuntini M, Campanacci L, Fabbri N, Pignotti E, Wuyts W, Sangiorgi L. Genotype-phenotype correlation study in 529 patients with multiple hereditary exostoses: identification of "protective" and "risk" factors. J Bone Joint Surg Am. 2011 Dec 21;93(24):2294-302. doi: 10.2106/JBJS.J.00949. PMID 22258776
- [Background] Schmale GA, Conrad EU 3rd, Raskind WH. The natural history of hereditary multiple exostoses. J Bone Joint Surg Am. 1994 Jul;76(7):986-92. doi: 10.2106/00004623-199407000-00005. PMID 8027127
- [Background] Pacifici M. Hereditary Multiple Exostoses: New Insights into Pathogenesis, Clinical Complications, and Potential Treatments. Curr Osteoporos Rep. 2017 Jun;15(3):142-152. doi: 10.1007/s11914-017-0355-2. PMID 28466453
- [Background] Vink GR, White SJ, Gabelic S, Hogendoorn PC, Breuning MH, Bakker E. Mutation screening of EXT1 and EXT2 by direct sequence analysis and MLPA in patients with multiple osteochondromas: splice site mutations and exonic deletions account for more than half of the mutations. Eur J Hum Genet. 2005 Apr;13(4):470-4. doi: 10.1038/sj.ejhg.5201343. PMID 15586175
- [Background] White SJ, Vink GR, Kriek M, Wuyts W, Schouten J, Bakker B, Breuning MH, den Dunnen JT. Two-color multiplex ligation-dependent probe amplification: detecting genomic rearrangements in hereditary multiple exostoses. Hum Mutat. 2004 Jul;24(1):86-92. doi: 10.1002/humu.20054. PMID 15221792
- [Background] Wuyts W, Van Hul W. Molecular basis of multiple exostoses: mutations in the EXT1 and EXT2 genes. Hum Mutat. 2000;15(3):220-7. doi: 10.1002/(SICI)1098-1004(200003)15:33.0.CO;2-K. PMID 10679937
- [Background] Darilek S, Wicklund C, Novy D, Scott A, Gambello M, Johnston D, Hecht J. Hereditary multiple exostosis and pain. J Pediatr Orthop. 2005 May-Jun;25(3):369-76. doi: 10.1097/01.bpo.0000150813.18673.ad. PMID 15832158
- [Background] Cacciari E, Milani S, Balsamo A, Spada E, Bona G, Cavallo L, Cerutti F, Gargantini L, Greggio N, Tonini G, Cicognani A. Italian cross-sectional growth charts for height, weight and BMI (2 to 20 yr). J Endocrinol Invest. 2006 Jul-Aug;29(7):581-93. doi: 10.1007/BF03344156. PMID 16957405
- [Background] Cacciari E, Milani S, Balsamo A, Dammacco F, De Luca F, Chiarelli F, Pasquino AM, Tonini G, Vanelli M. Italian cross-sectional growth charts for height, weight and BMI (6-20 y). Eur J Clin Nutr. 2002 Feb;56(2):171-80. doi: 10.1038/sj.ejcn.1601314. PMID 11857051
- [Background] Porter DE, Lonie L, Fraser M, Dobson-Stone C, Porter JR, Monaco AP, Simpson AH. Severity of disease and risk of malignant change in hereditary multiple exostoses. A genotype-phenotype study. J Bone Joint Surg Br. 2004 Sep;86(7):1041-6. doi: 10.1302/0301-620x.86b7.14815. PMID 15446535
- [Background] Goud AL, de Lange J, Scholtes VA, Bulstra SK, Ham SJ. Pain, physical and social functioning, and quality of life in individuals with multiple hereditary exostoses in The Netherlands: a national cohort study. J Bone Joint Surg Am. 2012 Jun 6;94(11):1013-20. doi: 10.2106/JBJS.K.00406. PMID 22637207
- [Background] D'Ambrosi R, Ragone V, Caldarini C, Serra N, Usuelli FG, Facchini RM. The impact of hereditary multiple exostoses on quality of life, satisfaction, global health status, and pain. Arch Orthop Trauma Surg. 2017 Feb;137(2):209-215. doi: 10.1007/s00402-016-2608-4. Epub 2016 Dec 8. PMID 27933382
- See also: Institutional webpage of Registries For Rare Hereditary Diseases — https://www.ior.it/en/curarsi-al-rizzoli/registries-rare-hereditary-diseases